CLINICAL TRIAL: NCT00613379
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study of PRO 140 by Intravenous Administration in Adult Subjects With Human Immunodeficiency Virus Type 1 Infection
Brief Title: PRO 140 by IV Administration in Adults With HIV-1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO 140 2301; 1U19AI066329 (NIH)
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: HIV Infections
Keywords: HIV; treatment naïve
MeSH Terms: conditions — HIV Infections | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): 10 mg/kg PRO 140, one IV dose (N=10)
  Interventions: Drug: PRO 140
- Arm 2 (Experimental): 5 mg/kg PRO 140, one IV dose (N=10)
  Interventions: Drug: PRO 140
- Arm 3 (Placebo Comparator): Placebo, one IV dose (N=10)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRO 140 — 10 mg/kg PRO 140, one IV dose (N=10)
  Arms: Arm 1
Drug: PRO 140 — 5 mg/kg PRO 140, one IV dose (N=10)
  Arms: Arm 2
Drug: Placebo — PBO, one IV dose (N=10)
  Arms: Arm 3

SUMMARY:
The purpose of this study is:

1. To assess and characterize the PK and PD of PRO 140 administered IV
2. To assess the antiviral activity of PRO 140
3. To assess the safety and tolerability of PRO 140

ELIGIBILITY:
Inclusion Criteria:

1. Males & females, age ≥ 18 years (or minimum adult age as determined by local regulatory authorities)
2. Screening plasma HIV-1 RNA ≥ 5,000 copies/mL
3. CD4+ T-lymphocyte cell count ≥ 300 cells/mm3 and no documented count < or = 250 cells/mm3
4. Has not taken any anti-retroviral therapy (ART) w/in 12 wks of Early Screening Visit
5. Exclusive CCR5-tropic virus as determined by Trofile™ Assay at Early Screening Visit
6. Clinically normal or "not clinically significant (NCS)" resting electrocardiogram
7. Women of reproductive potential must have a negative serum pregnancy test at Late Screening Visit & a negative urine pregnancy test w/in 72 hrs prior to first dose of study medication, & be non-lactating. Male & female subjects must agree not to participate in a conception process from Early Screening Visit through Day 59.

Exclusion Criteria:

1. CXCR4 tropic virus or dual/mixed tropic (R5X4) virus determined by the Trofile™ Assay.
2. Females who are pregnant, lactating or breastfeeding, or who plan to become pregnant during the study.
3. History of active hepatitis within the previous 24 wks
4. Prior use of any entry, attachment, CCR5 co-receptor or fusion inhibitor, experimental or approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Morris, MD, PhD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc, Tarrytown, New York, United States

REFERENCES:
- See also: Former Sponsor website — http://www.progenics.com
- See also: Sponsor Website — http://www.cytodyn.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from December 2007 to August 2008
Pre-assignment Details: Subjects screened up to 12 weeks
Groups:
- Arm 3: PBO, one IV dose (N=10)
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 10 | 10 | 11
Completed | 10 | 10 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 11 | 31
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (10.17) | 42 (9.88) | 38 (11.65) | 40.7 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 11 | 31
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change in Viral Load Following Initiation of Treatment.
Description: The primary end point was the maximum change from baseline in viral load following initiation of treatment, defined as HIV-1 copies/mL, measured by the Roche Amplicor HIV-1 Monitor UltraSensitive™ Test (lower limit of detection [LLD] = 48 copies/mL).
Time Frame: 59 days
Population: All randomized subjects who received one dose of study drug were considered intent-to-treat (ITT) subjects and were analyzed for efficacy.
Measure: Mean (Standard Error); unit: Log10copies HIV-1 RNA/mL
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 10 | 10 | 11
Log10copies HIV-1 RNA/mL | -1.67 (0.639) | -1.83 (0.229) | -0.32 (0.244)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 8/10 | 7/10 | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=10) | Arm 2 (N=10) | Arm 3 (N=11)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (3) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral hairy leukoplakia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Blood amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Echocardiogram normal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
QRS axis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Syphilis test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Physical assault (Social circumstances) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Because the study is a multicenter study, the PI(s) can only publish after the aggregate results of all investigators and institutions participating in the study have been published, and the proposed publication is reviewed by Progenics. In the event that Progenics does not publish the results of the study within eighteen months from availability of final study analysis, the PI can publish provided that the proposed publication is reviewed by Progenics.